CLINICAL TRIAL: NCT02638129
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 4 Study to Assess the Effect of Naltrexone Hydrochloride and Bupropion Hydrochloride Extended Release Combination on the Occurrence of Major Adverse Cardiovascular Events in Overweight and Obese Subjects With Cardiovascular Disease
Brief Title: Naltrexone/Bupropion Cardiovascular Outcomes Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Orexigen Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NaltrexBuprop-4001; U1111-1169-1350 (Registry Identifier: WHO)
Record Dates: First submitted 2015-12-18; First posted 2015-12-22 (Estimated); Results first posted 2017-02-27 (Actual); Last update posted 2017-02-27 (Actual); Status verified 2016-10

CONDITIONS: Obesity; Cardiovascular Diseases
Keywords: Drug therapy
MeSH Terms: conditions — Obesity; Cardiovascular Diseases | interventions — bupropion hydrochloride, naltrexone hydrochoride drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Lead-In: Naltrexone/Bupropion + Placebo (Other): Naltrexone hydrochloride (HCl) 8 mg/bupropion HCl 90 mg extended release (ER) combination tablets, orally, once daily for 1 week, followed by naltrexone/bupropion placebo-matching tablets, orally, once daily for 1 week. Participants who tolerate the naltrexone/bupropion treatment and comply with taking the study medication during the Lead-In Period will be randomized to the Double-Blind Treatment Period.
  Interventions: Drug: Naltrexone HCl/Bupropion HCl ER; Drug: Placebo
- Lead-In: Placebo + Naltrexone/Bupropion (Other): Naltrexone/bupropion placebo-matching tablets, orally, once daily, for 1 week, followed by naltrexone HCl 8 mg/bupropion HCl 90 mg ER combination tablets, orally, once daily, for 1 week. Participants who tolerate the naltrexone/bupropion treatment and comply with taking the study medication during the Lead-In Period will be randomized to the Double-Blind Treatment Period.
  Interventions: Drug: Naltrexone HCl/Bupropion HCl ER; Drug: Placebo
- Naltrexone/Bupropion (Active Comparator): Naltrexone HCl 8 mg/bupropion HCl 90 mg ER combination tablets, orally, one tablet, in the morning (AM), daily, for 1 week, followed by naltrexone HCl 8 mg/bupropion HCl 90 mg ER combination tablets, orally, one tablet in the AM and one in the evening (PM), daily, for 1 week, followed by naltrexone HCl 8 mg/bupropion HCl 90 mg ER combination tablets, orally, two tablets in the AM and one in the PM, daily, for 1 week, followed by naltrexone HCl 8 mg/bupropion HCl 90 mg ER combination tablets, orally, two tablets in the AM and two in the PM, daily, for up to 6 years.
  Interventions: Drug: Naltrexone HCl/Bupropion HCl ER
- Placebo (Placebo Comparator): Naltrexone/bupropion placebo-matching tablets, orally, one tablet in the AM, daily, for 1 week, followed by naltrexone/bupropion placebo-matching tablets, orally, one tablet in the AM and one in the PM, daily, for 1 week, followed by naltrexone/bupropion placebo-matching tablets, orally, two tablets in the AM and one in the PM, daily, for 1 week, followed by naltrexone/bupropion placebo-matching tablets, orally, two tablets in the AM and two in the PM, daily, for up to 6 years.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone HCl/Bupropion HCl ER — Naltrexone HCl 8 mg/bupropion HCl 90 mg ER combination tablets
  Other Names: Contrave
  Arms: Lead-In: Naltrexone/Bupropion + Placebo; Lead-In: Placebo + Naltrexone/Bupropion; Naltrexone/Bupropion
Drug: Placebo — Naltrexone HCl/bupropion HCl placebo-matching tablets
  Arms: Lead-In: Naltrexone/Bupropion + Placebo; Lead-In: Placebo + Naltrexone/Bupropion; Placebo

SUMMARY:
The purpose of this study is to evaluate cardiovascular (CV) safety of naltrexone hydrochloride (HCl) and bupropion HCl extended release combination (NB) compared with placebo and rule out excess risk of major adverse cardiovascular events (MACE) when given in combination with standard of care in overweight and obese participants with documented history of CV disease.

DETAILED DESCRIPTION:
The drug being evaluated in this study is naltrexone hydrochloride (HCl) and bupropion HCl extended release combination (NB). NB is being evaluated in this study to rule out excess cardiovascular risk. This study will evaluate the occurrence of major adverse CV events in participants who take NB compared with placebo given in combination with standard of care in overweight and obese participants with documented history of CV disease.

The study will enroll approximately 8800 patients. After a 2-week lead-in period evaluating tolerance to NB (participants were randomly assigned in a 1:1 ratio to 1 week of NB [1 tablet per day] followed by 1 week of placebo [1 tablet per day] or 1 week of placebo followed by 1 week of NB), participants will be randomly assigned to one of two treatment groups in a 1:1 ratio, which will remain undisclosed to the patient, study site personnel, and investigator/study physician during the study (unless there is an urgent medical need):

* Naltrexone HCl 8 mg/bupropion 90 mg extended release combination tablets
* Placebo (dummy inactive pill) - this is a tablet that looks like the study drug but has no active ingredient

All participants will be asked to take tablet(s) in the AM and PM at the same time each day throughout the study.

This multi-center trial will be conducted in the United States. The overall time to participate in this study is up to 6 years. Participants will make multiple visits to the clinic, and will be contacted by telephone 30 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.

2. Participant signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.

3. Has body mass index (BMI) ≥27.0 kg/m^2 at Screening. 4. Is male or female and aged ≥18 years at Screening. 5. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent through 12 weeks after the last dose of study medication.

6. Participant meets at least 1 the following categories of cardiovascular (CV) disease (a-c):

1. Documented coronary artery disease (at least 1 of the following 2 criteria must be satisfied):

   1. A documented history of myocardial infarction (MI) occurring greater than 3 months prior to Screening.
   2. History of coronary revascularization with at least 1 of the following:

      1. Coronary artery bypass graft surgery occurring greater than 3 months prior to Screening.
      2. Percutaneous coronary intervention (PCI) occurring greater than 3 months prior to Screening.
2. Documented peripheral arterial disease (at least 1 of the following 3 criteria must be satisfied):

   1. Current intermittent claudication or verified ischemic ulcer(s) together with documented ankle-brachial index ≤0.85.
   2. History of previous vascular intervention for intermittent claudication or resting limb ischemia greater than 3 months prior to Screening (example: amputation for arterial disease, peripheral bypass, or history of angioplasty/stenting).
   3. History of symptomatic carotid artery disease (requiring revascularization with carotid endarterectomy or stenting) greater than 3 months prior to Screening or ≥50% stenosis on at least one carotid artery documented by duplex ultrasonography, magnetic resonance angiography, computed tomographic angiography, or catheter-based contrast angiography.
3. Documented cerebrovascular disease (at least 1 of the following 2 criteria must be satisfied):

   1. A history of transient ischemic attack confirmed by a neurologist greater than 3 months prior to Screening and clinically and neurologically stable at Screening.
   2. A history of ischemic stroke (with a Modified Rankin Scale Score ≤3) greater than 3 months prior to Screening and clinically and neurologically stable at Screening.

Exclusion Criteria:

1. Has received any investigational compound or investigational device within 3 months prior to Screening.
2. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
3. Has had an MI or unstable angina within 3 months of Screening.
4. Has planned bariatric surgery, cardiac surgery, coronary revascularization, or peripheral artery revascularization.
5. Has history of bariatric surgery (eg, Roux-en-Y gastric bypass, duodenal switch, or sleeve gastrectomy).
6. Has had a procedure for weight loss other than bariatric surgery (eg, gastric banding or any other devices that maybe used in obesity treatment) within past 12 months prior to Screening.
7. Has a history of hypersensitivity or allergies to any component of naltrexone hydrochloride (HCl) and bupropion HCl extended release combination (NB) or excipients.
8. Has a history of cancer that has been in remission for <5 years prior to Screening. A history of basal cell carcinoma or Stage 1 squamous cell carcinoma of the skin is allowed.
9. Is hemodynamically unstable, including severe heart failure (New York Heart Association Class IV) at Screening.
10. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 2 years prior to Screening.
11. Has been randomized into a previous NB (Contrave) study or has been exposed to commercially available NB (Contrave) for any period of time prior to Screening.
12. Is taking excluded medications within 28 days of Screening.
13. Has uncontrolled hypertension defined by systolic blood pressure (SBP) ≥160 mm Hg and/or ≥100 mm Hg diastolic blood pressure (DBP) on the average of two seated blood pressure measurements after being at rest at least 5 minutes, confirmed on 2 separate days during the Screening Period.
14. Has severe renal impairment defined by estimated glomerular filtration rate (eGFR) <30 ml/min/1.73 m^2 based on the Chronic Kidney Disease Epidemiology Collaboration equation (CKD-EPI) at Screening.
15. Has a clinical history of liver failure.
16. Has a known infection with human immunodeficiency virus that is being treated with ritonavir, lopinavir or efavirenz.
17. Has known acute hepatitis at Screening.
18. Has chronic use of opioids, defined as longer than 3 months prior to Screening.
19. Has a positive drug screen for cocaine, methamphetamine, methadone, opiates, oxycodone, phencyclidine, and propoxyphene at Screening. A positive screen for amphetamines, barbiturates, benzodiazepines, and cannabinoids is exclusionary if abuse or dependence is suspected.
20. Has a history of seizures (including febrile seizures), cranial trauma, or other conditions that predispose the participant to seizures.
21. Has a history of mania, history of or current diagnosis of bipolar disorder or current diagnosis of active psychosis, active bulimia or anorexia nervosa (binge eating disorder is not exclusionary).
22. Is at risk for suicide attempts based on the judgment of the investigator.
23. If female, the participant is pregnant (confirmed by laboratory testing at screening) or lactating or intending to become pregnant from signing the informed consent through 12 weeks after last dose of study medication; or intending to donate ova during such time period.
24. Has a history of severe ischemic stroke (with a Modified Rankin Scale Score ≥4).
25. Has any major illness or condition that, in the investigator's opinion, prohibits the participant from participating in the study or meeting the planned visit schedule.
26. Is unable to understand verbal or written English or any other language, for which a certified translation of the approved informed consent is available.

Additional exclusion criteria to be assessed at Visit3 prior to Randomization:

1. Participant takes <75% or >125% of the Lead-in study medication.
2. Participant discontinues study medication treatment or has a known major adverse cardiovascular events (MACE) reported by investigator during the Double-Blind Lead-in Period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (139):
- United States (139):
  - Alexander City, Alabama
  - Auburn, Alabama
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Campe Verde, Arizona
  - Chandler, Arizona
  - Cottonwood, Arizona
  - Fountain Hills, Arizona
  - Mesa, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Fayetteville, Arkansas
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Arvin, California
  - Bakersfield, California
  - Chino, California
  - Downey, California
  - El Cajon, California
  - Los Alamitos, California
  - Los Angeles, California
  - Pomona, California
  - Sacramento, California
  - Santa Ana, California
  - Santa Monica, California
  - Denver, Colorado
  - New London, Connecticut
  - Stamford, Connecticut
  - Trumbull, Connecticut
  - Waterbury, Connecticut
  - Wilmington, Delaware
  - Boca Raton, Florida
  - Bradenton, Florida
  - Brandon, Florida
  - Brooksville, Florida
  - Coral Springs, Florida
  - Cutler Bay, Florida
  - Daytona Beach, Florida
  - Hialeah, Florida
  - Inverness, Florida
  - Jacksonville Beach, Florida
  - Lake Worth, Florida
  - Largo, Florida
  - Miami Lakes, Florida
  - Orlando, Florida
  - Palm Harbor, Florida
  - Pembroke Pines, Florida
  - Ponte Vedra Beach, Florida
  - Sarasota, Florida
  - Stuart, Florida
  - Atlanta, Georgia
  - Duluth, Georgia
  - Savannah, Georgia
  - Honolulu, Hawaii
  - Pocatello, Idaho
  - Blue Island, Illinois
  - Chicago, Illinois
  - Evanston, Illinois
  - Gurnee, Illinois
  - Rock Island, Illinois
  - Evansville, Indiana
  - Topeka, Kansas
  - Louisville, Kentucky
  - Owensboro, Kentucky
  - Baton Rouge, Louisiana
  - Bossier City, Louisiana
  - Lake Charles, Louisiana
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Catonsville, Maryland
  - Bay City, Michigan
  - Saginaw, Michigan
  - Port Gibson, Mississippi
  - Hazelwood, Missouri
  - Great Falls, Montana
  - Las Vegas, Nevada
  - Linden, New Jersey
  - Moorestown, New Jersey
  - Albuquerque, New Mexico
  - Endwell, New York
  - Great Neck, New York
  - Mineola, New York
  - New York, New York
  - Saratoga Springs, New York
  - Staten Island, New York
  - Asheville, North Carolina
  - Cary, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Greenville, North Carolina
  - Hickory, North Carolina
  - Morehead City, North Carolina
  - Raleigh, North Carolina
  - Rocky Mount, North Carolina
  - Salisbury, North Carolina
  - Winston-Salem, North Carolina
  - Canton, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Perrysburg, Ohio
  - Sandusky, Ohio
  - Willoughby, Ohio
  - Altoona, Pennsylvania
  - Camp Hill, Pennsylvania
  - Doylestown, Pennsylvania
  - Lansdale, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Smithfield, Pennsylvania
  - Yardley, Pennsylvania
  - Charleston, South Carolina
  - Moncks Corner, South Carolina
  - Mt. Pleasant, South Carolina
  - Simpsonville, South Carolina
  - Bristol, Tennessee
  - Jackson, Tennessee
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Arlington, Texas
  - Dallas, Texas
  - Houston, Texas
  - Katy, Texas
  - Kingwood, Texas
  - Palestine, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Bountiful, Utah
  - Murray, Utah
  - Ogden, Utah
  - Orem, Utah
  - South Ogden, Utah
  - West Jordan, Utah
  - West, Utah
  - Richmond, Virginia
  - Roanoke, Virginia
  - Virginia Beach, Virginia
  - Port Orchard, Washington
  - Charleston, West Virginia
  - Kenosha, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sixty-seven (67) participants randomized into the double-blind lead-in period (Enrolled Set), while 58 participants were randomized into the double-blind treatment period (Full Analysis Set).
Period: Overall Study
Arm/Group | Naltrexone/Bupropion | Placebo
Started | 28 | 30
Completed | 0 | 0
Not Completed | 28 | 30
Not completed — Study terminated | 28 | 30

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone/Bupropion | Placebo | Total
Number analyzed (Participants) | 28 | 30 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 14 | 33
  >=65 years | 9 | 16 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (9.29) | 65.5 (7.04) | 63.5 (8.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 22 | 21 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 26 | 28 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 7 | 7 | 14
  White | 19 | 23 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time From Treatment Period Randomization to the First Confirmed Occurrence of Major Adverse Cardiovascular Events (MACE)
Description: MACE are defined as cardiovascular death, nonfatal myocardial infarction and nonfatal stroke.
Time Frame: Day 1 to first confirmed occurrence of MACE (up to 6 years)
Population: The trial was prematurely terminated. Due to the short trial duration and as a result of very limited participant follow-up, insufficient data was collected (or did not exist) to allow for a statistical analysis as described in the protocol. The necessary and sufficient data to conduct the primary and secondary analyses was not available.
Arm/Group | Naltrexone/Bupropion | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Time From Treatment Period Randomization to the First Confirmed Occurrence of Extended Major Adverse Cardiovascular Events (MACE)
Description: Extended MACE defined as cardiovascular death, nonfatal myocardial infarction, nonfatal stroke, and unstable angina requiring hospitalization.
Time Frame: Day 1 to first confirmed occurrence of extended MACE (up to 6 years)
Population: as for outcome 1
Arm/Group | Naltrexone/Bupropion | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time From Treatment Period Randomization to the Occurrence of All-Cause Death
Time Frame: Day 1 to the occurrence of all-cause death (up to 6 years)
Population: as for outcome 1
Arm/Group | Naltrexone/Bupropion | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Time From Treatment Period Randomization to the Occurrence of Cardiovascular Death
Time Frame: Day 1 to the occurrence of cardiovascular death (up to 6 years)
Population: as for outcome 1
Arm/Group | Naltrexone/Bupropion | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Study was terminated with the maximum subject duration on study of 13.1 weeks.
Description: Study did not collect all non-serious adverse events. Safety data collection was limited to adverse events leading to discontinuation of study medication, special interest adverse events, and serious adverse events. All recorded non-serious AEs and SAEs are reported in the tables.
Arm/Group | Naltrexone/Bupropion | Placebo
Serious Adverse Events (participants affected / at risk) | 2/28 | 2/30
Other Adverse Events (participants affected / at risk) | 1/28 | 2/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naltrexone/Bupropion (N=28) | Placebo (N=30)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Brain stem stroke (Nervous system disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naltrexone/Bupropion (N=28) | Placebo (N=30)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
As this study was prematurely terminated, analysis of the primary and secondary outcome measures was not performed and analysis of safety was limited in scope.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If not already published by Sponsor as part of a multi-center publication, 24 months after conclusion, abandonment or termination of the study or notification that there will be no such multi-center publication, PI may publish the results for PI's study center individually. Prior to such publication, PI must provide Sponsor with at least 60 days to review and comment on the proposed publication. Sponsor may delay publication for up to an additional 6 month period to file for patent protection.